CLINICAL TRIAL: NCT06531200
Title: Building of Prognosis Model for Patients With Cirrhosis Based on Sarcopenia in Assessment With the Technology of Deep Learning
Brief Title: Building of Prognosis Model for Patients With Cirrhosis Based on Sarcopenia Assessed by Deep Learning
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Huang Rui, Principal Investigator, Peking University People's Hospital
Other Study IDs: 2023PHB214-001
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Cirrhosis, Liver; Sarcopenia
Keywords: deep learning; prognosis; sarcopenia; myosteatosis
MeSH Terms: conditions — Liver Cirrhosis; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop and validate a fully automated imaging deep learning platform for the evaluation of sarcopenia in liver cirrhosis. Based on this model, a new prognostic model for liver cirrhosis incorporating imaging biomarkers such as sarcopenia will be constructed, and its predictive performance will be validated.

DETAILED DESCRIPTION:
The goal of this observational study is to collect clinical and abdominal imaging data of patients with liver cirrhosis. The collected imaging data will be used as a model development set to develop, test, and internally validate a fully automated imaging deep learning platform for the evaluation of sarcopenia in liver cirrhosis. Subsequently, relevant data from patients with liver cirrhosis at other centers will be collected and used as an external validation dataset. The model will be externally validated by abdominal radiology experts. Furthermore, we will include sociodemographic information, clinical data, imaging data, and clinical outcomes of the aforementioned liver cirrhosis patients to predict the prognosis of these patients using the established model. This model will be used to construct a new prognostic model for liver cirrhosis incorporating imaging biomarkers such as sarcopenia, and its predictive performance will be validated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of liver cirrhosis, meeting at least one of the following criteria:
* Clinical diagnosis: ICD-10-CM codes K74.100 and K74.607 from our hospital's electronic medical record system
* Liver biopsy pathology or a combination of clinical, laboratory, and imaging examinations confirming liver cirrhosis: Pathological biopsy criteria: fibrosis bridging between lobules leading to lobular structural disarray, nodular regeneration of hepatocytes, formation of pseudo-lobules
* Laboratory tests: the presence of at least 2 of the following 4 abnormal indicators suggesting liver cirrhosis:
* a) Platelet count < 100×10^9/L, with no other explainable cause;
* b) Serum albumin < 35g/L, excluding malnutrition or kidney disease as other causes;
* c) International normalized ratio (INR) > 1.3 or prolonged prothrombin time (PT) (after discontinuation of thrombolytic or anticoagulant drugs for more than 7 days);
* d)Aspartate aminotransferase to platelet ratio index (APRI) > 2.
* Availability of high-quality L3-level CT images

Exclusion Criteria:

* Incomplete sociodemographic, laboratory, or imaging data
* Diagnosed or highly suspected malignancy
* Severe chronic kidney disease, respiratory insufficiency, cardiovascular diseases, etc.
* Neurological diseases and muscular degenerative diseases
* Hyperthyroidism, hypothyroidism, tuberculosis, or any other diseases that may affect basal metabolism
* Diseases or conditions causing malabsorption of intestinal nutrients, such as inflammatory bowel disease or gastrointestinal surgery
* Treatment with glucocorticoids or immunosuppressants
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adults diagnosed with liver cirrhosis based on clinical criteria, liver biopsy confirming cirrhosis, or specific laboratory abnormalities (e.g., low platelet count, low serum albumin, high INR, or elevated APRI). Additionally, high-quality L3-level CT images must be available for each patient. Patients are excluded if they have incomplete data, a diagnosis or suspicion of malignancy, severe chronic diseases (such as kidney, respiratory, or cardiovascular conditions), neurological or muscular degenerative diseases, metabolic disorders (like thyroid diseases or tuberculosis), malabsorption conditions, or if they are undergoing treatment with glucocorticoids or immunosuppressants. Pregnant or lactating women are also excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver-related mortality | As of December 31, 2025
  Causes of liver disease-related mortality include: Hepatitis B virus infection, hepatitis C virus infection, alcohol-induced or toxic liver disease; complications related to liver cirrhosis: ascites or pleural effusion, esophagogastric variceal bleeding, spontaneous bacterial peritonitis or related infections, hepatic encephalopathy or other neuropsychiatric syndromes based on metabolic disorders, hepatorenal syndrome, hepatopulmonary syndrome; liver failure; hepatocellular carcinoma; death or liver transplantation.

SECONDARY OUTCOMES:
All-cause Mortality | As of December 31, 2025
  Deaths caused by all reasons, including but not limited to those related to liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Rui Huang, Dr., Principal Investigator — Rui Huang, Dr. PekignUnviersity People's Hospital

REFERENCES:
- [Background] Huang DQ, Terrault NA, Tacke F, Gluud LL, Arrese M, Bugianesi E, Loomba R. Global epidemiology of cirrhosis - aetiology, trends and predictions. Nat Rev Gastroenterol Hepatol. 2023 Jun;20(6):388-398. doi: 10.1038/s41575-023-00759-2. Epub 2023 Mar 28. PMID 36977794
- [Background] Zeng X, Shi ZW, Yu JJ, Wang LF, Luo YY, Jin SM, Zhang LY, Tan W, Shi PM, Yu H, Zhang CQ, Xie WF. Sarcopenia as a prognostic predictor of liver cirrhosis: a multicentre study in China. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1948-1958. doi: 10.1002/jcsm.12797. Epub 2021 Sep 14. PMID 34520115
- [Background] Desai AP, Mohan P, Nokes B, Sheth D, Knapp S, Boustani M, Chalasani N, Fallon MB, Calhoun EA. Increasing Economic Burden in Hospitalized Patients With Cirrhosis: Analysis of a National Database. Clin Transl Gastroenterol. 2019 Jul;10(7):e00062. doi: 10.14309/ctg.0000000000000062. PMID 31343469
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Damluji AA, Alfaraidhy M, AlHajri N, Rohant NN, Kumar M, Al Malouf C, Bahrainy S, Ji Kwak M, Batchelor WB, Forman DE, Rich MW, Kirkpatrick J, Krishnaswami A, Alexander KP, Gerstenblith G, Cawthon P, deFilippi CR, Goyal P. Sarcopenia and Cardiovascular Diseases. Circulation. 2023 May 16;147(20):1534-1553. doi: 10.1161/CIRCULATIONAHA.123.064071. Epub 2023 May 15. PMID 37186680
- [Background] Sinn DH, Kang D, Kang M, Guallar E, Hong YS, Lee KH, Park J, Cho J, Gwak GY. Nonalcoholic fatty liver disease and accelerated loss of skeletal muscle mass: A longitudinal cohort study. Hepatology. 2022 Dec;76(6):1746-1754. doi: 10.1002/hep.32578. Epub 2022 Jun 10. PMID 35588190
- [Background] Han E, Lee YH, Kim BK, Park JY, Kim DY, Ahn SH, Lee BW, Kang ES, Cha BS, Han KH, Kim SU. Sarcopenia is associated with the risk of significant liver fibrosis in metabolically unhealthy subjects with chronic hepatitis B. Aliment Pharmacol Ther. 2018 Aug;48(3):300-312. doi: 10.1111/apt.14843. Epub 2018 Jun 19. PMID 29920701
- [Background] Davuluri G, Welch N, Sekar J, Gangadhariah M, Alsabbagh Alchirazi K, Mohan ML, Kumar A, Kant S, Thapaliya S, Stine M, McMullen MR, McCullough RL, Stark GR, Nagy LE, Naga Prasad SV, Dasarathy S. Activated Protein Phosphatase 2A Disrupts Nutrient Sensing Balance Between Mechanistic Target of Rapamycin Complex 1 and Adenosine Monophosphate-Activated Protein Kinase, Causing Sarcopenia in Alcohol-Associated Liver Disease. Hepatology. 2021 May;73(5):1892-1908. doi: 10.1002/hep.31524. Epub 2021 Apr 20. PMID 32799332
- [Background] Shafaat O, Liu Y, Jackson KR, Motter JD, Boyarsky BJ, Latif MA, Yuan F, Khalil A, King EA, Zaheer A, Summers RM, Segev DL, McAdams-DeMarco M, Weiss CR. Association between Abdominal CT Measurements of Body Composition before Deceased Donor Liver Transplant with Posttransplant Outcomes. Radiology. 2023 Mar;306(3):e212403. doi: 10.1148/radiol.212403. Epub 2022 Oct 25. PMID 36283115
- [Background] Dasarathy S, Merli M. Sarcopenia from mechanism to diagnosis and treatment in liver disease. J Hepatol. 2016 Dec;65(6):1232-1244. doi: 10.1016/j.jhep.2016.07.040. Epub 2016 Aug 8. PMID 27515775
- [Background] Kang SH, Jeong WK, Baik SK, Cha SH, Kim MY. Impact of sarcopenia on prognostic value of cirrhosis: going beyond the hepatic venous pressure gradient and MELD score. J Cachexia Sarcopenia Muscle. 2018 Oct;9(5):860-870. doi: 10.1002/jcsm.12333. PMID 30371017
- [Background] van Vugt JLA, Alferink LJM, Buettner S, Gaspersz MP, Bot D, Darwish Murad S, Feshtali S, van Ooijen PMA, Polak WG, Porte RJ, van Hoek B, van den Berg AP, Metselaar HJ, IJzermans JNM. A model including sarcopenia surpasses the MELD score in predicting waiting list mortality in cirrhotic liver transplant candidates: A competing risk analysis in a national cohort. J Hepatol. 2018 Apr;68(4):707-714. doi: 10.1016/j.jhep.2017.11.030. Epub 2017 Dec 6. PMID 29221886
- [Background] Bhanji RA, Moctezuma-Velazquez C, Duarte-Rojo A, Ebadi M, Ghosh S, Rose C, Montano-Loza AJ. Myosteatosis and sarcopenia are associated with hepatic encephalopathy in patients with cirrhosis. Hepatol Int. 2018 Jul;12(4):377-386. doi: 10.1007/s12072-018-9875-9. Epub 2018 Jun 7. PMID 29881992
- [Background] Tosato M, Marzetti E, Cesari M, Savera G, Miller RR, Bernabei R, Landi F, Calvani R. Measurement of muscle mass in sarcopenia: from imaging to biochemical markers. Aging Clin Exp Res. 2017 Feb;29(1):19-27. doi: 10.1007/s40520-016-0717-0. Epub 2017 Feb 7. PMID 28176249
- [Background] Prado CM, Heymsfield SB. Lean tissue imaging: a new era for nutritional assessment and intervention. JPEN J Parenter Enteral Nutr. 2014 Nov;38(8):940-53. doi: 10.1177/0148607114550189. Epub 2014 Sep 19. PMID 25239112
- [Background] Chianca V, Albano D, Messina C, Gitto S, Ruffo G, Guarino S, Del Grande F, Sconfienza LM. Sarcopenia: imaging assessment and clinical application. Abdom Radiol (NY). 2022 Sep;47(9):3205-3216. doi: 10.1007/s00261-021-03294-3. Epub 2021 Oct 23. PMID 34687326
- [Background] Pillen S, van Alfen N. Skeletal muscle ultrasound. Neurol Res. 2011 Dec;33(10):1016-24. doi: 10.1179/1743132811Y.0000000010. PMID 22196753
- [Background] Sconfienza LM. Sarcopenia: ultrasound today, smartphones tomorrow? Eur Radiol. 2019 Jan;29(1):1-2. doi: 10.1007/s00330-018-5833-0. Epub 2018 Nov 12. No abstract available. PMID 30421017
- [Background] Lenchik L, Boutin RD. Sarcopenia: Beyond Muscle Atrophy and into the New Frontiers of Opportunistic Imaging, Precision Medicine, and Machine Learning. Semin Musculoskelet Radiol. 2018 Jul;22(3):307-322. doi: 10.1055/s-0038-1641573. Epub 2018 May 23. PMID 29791959
- [Background] Albano D, Chianca V, Tormenta S, Migliore A, Sconfienza LM. Old and new evidence concerning the crucial role of ultrasound in guiding intra-articular injections. Skeletal Radiol. 2017 Jul;46(7):963-964. doi: 10.1007/s00256-017-2644-3. Epub 2017 Apr 10. No abstract available. PMID 28396961
- [Background] Carey EJ, Lai JC, Sonnenday C, Tapper EB, Tandon P, Duarte-Rojo A, Dunn MA, Tsien C, Kallwitz ER, Ng V, Dasarathy S, Kappus M, Bashir MR, Montano-Loza AJ. A North American Expert Opinion Statement on Sarcopenia in Liver Transplantation. Hepatology. 2019 Nov;70(5):1816-1829. doi: 10.1002/hep.30828. Epub 2019 Aug 19. PMID 31220351
- [Background] Nishikawa H, Shiraki M, Hiramatsu A, Moriya K, Hino K, Nishiguchi S. Japan Society of Hepatology guidelines for sarcopenia in liver disease (1st edition): Recommendation from the working group for creation of sarcopenia assessment criteria. Hepatol Res. 2016 Sep;46(10):951-63. doi: 10.1111/hepr.12774. PMID 27481650
- [Background] Moon SW, Choi JS, Lee SH, Jung KS, Jung JY, Kang YA, Park MS, Kim YS, Chang J, Kim SY. Thoracic skeletal muscle quantification: low muscle mass is related with worse prognosis in idiopathic pulmonary fibrosis patients. Respir Res. 2019 Feb 15;20(1):35. doi: 10.1186/s12931-019-1001-6. PMID 30767787
- [Background] Tagliafico AS, Bignotti B, Torri L, Rossi F. Sarcopenia: how to measure, when and why. Radiol Med. 2022 Mar;127(3):228-237. doi: 10.1007/s11547-022-01450-3. Epub 2022 Jan 18. PMID 35041137
- [Background] Ye Z, Saraf A, Ravipati Y, Hoebers F, Catalano PJ, Zha Y, Zapaishchykova A, Likitlersuang J, Guthier C, Tishler RB, Schoenfeld JD, Margalit DN, Haddad RI, Mak RH, Naser M, Wahid KA, Sahlsten J, Jaskari J, Kaski K, Makitie AA, Fuller CD, Aerts HJWL, Kann BH. Development and Validation of an Automated Image-Based Deep Learning Platform for Sarcopenia Assessment in Head and Neck Cancer. JAMA Netw Open. 2023 Aug 1;6(8):e2328280. doi: 10.1001/jamanetworkopen.2023.28280. PMID 37561460
- [Background] Zhang H, Yin M, Liu Q, Ding F, Hou L, Deng Y, Cui T, Han Y, Pang W, Ye W, Yue J, He Y. Machine and deep learning-based clinical characteristics and laboratory markers for the prediction of sarcopenia. Chin Med J (Engl). 2023 Apr 20;136(8):967-973. doi: 10.1097/CM9.0000000000002633. Epub 2023 Apr 7. PMID 37098831
- [Background] Blanc-Durand P, Schiratti JB, Schutte K, Jehanno P, Herent P, Pigneur F, Lucidarme O, Benaceur Y, Sadate A, Luciani A, Ernst O, Rouchaud A, Creze M, Dallongeville A, Banaste N, Cadi M, Bousaid I, Lassau N, Jegou S. Abdominal musculature segmentation and surface prediction from CT using deep learning for sarcopenia assessment. Diagn Interv Imaging. 2020 Dec;101(12):789-794. doi: 10.1016/j.diii.2020.04.011. Epub 2020 May 22. PMID 32451309
- [Background] Gu S, Wang L, Han R, Liu X, Wang Y, Chen T, Zheng Z. Detection of sarcopenia using deep learning-based artificial intelligence body part measure system (AIBMS). Front Physiol. 2023 Jan 26;14:1092352. doi: 10.3389/fphys.2023.1092352. eCollection 2023. PMID 36776966
- [Background] Yi J, Shin Y, Hahn S, Lee YH. Deep learning based sarcopenia prediction from shear-wave ultrasonographic elastography and gray scale ultrasonography of rectus femoris muscle. Sci Rep. 2022 Mar 4;12(1):3596. doi: 10.1038/s41598-022-07683-6. PMID 35246589